CLINICAL TRIAL: NCT04379284
Title: Risks of COVID19 in the Pregnant Population
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Regan N. Theiler, Principal Investigator, Mayo Clinic
Other Study IDs: 20-003251
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: COVID19
Keywords: COVID19; Coronavirus; Pregnancy; Viral infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal specimens obtained at time of enrollment prior to delivery: blood, vaginal swab, anorectal swab. Breastmilk obtained before hospital discharge and again at six weeks postpartum if the mother is lactating.
  Neonatal specimens: placental tissue, fetal membrane roll, umbilical cord tissue, umbilical cord blood, and an anorectal swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women - positive COVID19 test: Pregnant women of any gestational age 8 weeks through delivery with a positive COVID19 test, with or without physical symptoms
  Interventions: Other: Biospecimen collection
- Pregnant women - negative or unknown COVID19 test: Pregnant women experiencing any respiratory or other physical symptoms of COVID19 at onset of labor, with negative or uncertain COVID19 test results
  Interventions: Other: Biospecimen collection

INTERVENTIONS:
Other: Biospecimen collection — Maternal blood, vaginal swab, and anorectal swab will be obtained at the time of enrollment prior to delivery. A sample of breastmilk before hospital discharge and again at six weeks postpartum will be obtained if the mother is lactating.
  Neonatal specimens collected following delivery will include placental tissue, fetal membrane roll, umbilical cord tissue, umbilical cord blood, and an anorectal swab.

SUMMARY:
It is unclear how COVID19 can be passed from mother to infant. The study investigators aim to collect maternal and neonatal samples from COVID19-infected pregnant women and compare them to pregnant women who have clinical indications for COVID 19 testing at the time of hospital admission but end up being COVID19 negative. Pregnant women who are either COVID19 positive or COVID19 negative with respiratory symptoms will be enrolled and followed during this study.

DETAILED DESCRIPTION:
The objectives are to understand the prevalence of maternal fetal transmission, risk factors and outcomes of a COVID19 positive pregnancy, and how the virus can be passed from mother to infant in the pregnant population at Mayo Clinic Rochester MN. Assessments will include the viral detection and viral load in maternal and fetal specimens collected from COVID19 positive mother-baby dyads, presence of maternal and fetal inflammatory markers in blood and tissues, anti-COVID IgG and IgM in maternal and neonatal blood, viral load and viral antigens in maternal and fetal specimens. placental gross and histopathologic changes in COVID19 infected mothers, stratified by gestational age and disease severity, compared to control samples.

.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18 - 45 years of age and their newborn infants
* Willing and able to provide written informed consent
* Planning to deliver at Mayo Clinic in Rochester, MN

Exclusion Criteria:

* Positive for HIV, HBV, or TB
* Delivery does not occur at Mayo Clinic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women testing positive for COVID19 at any time during their pregnancy after 8 weeks gestation, with or without physical symptoms. Pregnant women with respiratory or other physical symptoms of COVID19 and uncertain or negative COVID19 test results at the onset of labor.
  Infants of these women will be followed for outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of maternal fetal transmission of COVID19 | 12 months
  Standardized testing of maternal, placental, and neonatal specimens will be used to determine presence of current infection with SARS-CoV2. Clinical RT-PCR assays will be used to determine the presence of viral RNA in all specimens.

SECONDARY OUTCOMES:
Describe the outcomes of COVID19 positive pregnancies | 12 months
  Clinical data from prenatal, intrapartum, and postpartum care will be abstracted from maternal records and correlated with neonatal outcomes. Any complications will be characterized, with comparison to the non-COVID19 control group of patients. Statistical analysis will reveal characteristics and clinical outcomes that may be linked to COVID19 infection in pregnancy.
Understand the placental impact of COVID19 in pregnancy at various gestational ages | 12 months
  In addition to maternal and fetal infection, disease states related to placental dysfunction may be related to COVID19 infection in pregnancy. We will examine placenta and markers of placental function to assess for discernable consequences of maternal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Regan N Theiler, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing individual participant data

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials